CLINICAL TRIAL: NCT00268957
Title: A Randomized, Parallel, Open-Label Study to Compare Once Per Day Sevelamer Carbonate Powder Dosing With Three Times Per Day Sevelamer Hydrochloride Tablet Dosing in Chronic Kidney Disease Patients on Hemodialysis
Brief Title: Study to Compare Sevelamer Carbonate Powder to Sevelamer Hydrochloride Tablets in Patients With CKD on Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GD3-199-301
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Kidney Diseases; Chronic Renal Insufficiency; End-Stage Renal Disease
Keywords: Chronic; Hemodialysis; Kidney; Hyperphosphatemia; Chronic kidney disease; Chronic Renal Insufficiency
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic; Kidney Failure, Chronic; Bronchiolitis Obliterans Syndrome; Hyperphosphatemia | interventions — Sevelamer

ARMS (2):
- 1 (Experimental): sevelamer carbonate powder
  Interventions: Drug: Sevelamer carbonate (Renvela®)
- 2 (Active Comparator): Sevelamer hydrochloride
  Interventions: Drug: Sevelamer hydrochloride (Renagel®)

INTERVENTIONS:
Drug: Sevelamer carbonate (Renvela®) — sevelamer carbonate powder dosed once per day with largest meal
  Arms: 1
Drug: Sevelamer hydrochloride (Renagel®) — Sevelamer hydrochloride tablets dosed three times a day with meals
  Arms: 2

SUMMARY:
Approximately 207 patients with chronic kidney disease (CKD) on hemodialysis will be entered into this study at approximately 26 centers in the United States. This study aims to evaluate the safety and efficacy of sevelamer carbonate powder dosed once-a-day (QD) with the largest meal compared to sevelamer hydrochloride tablets dosed three-times-per-day (TID) with meals. The total length of participation is approximately 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* On three times per week hemodialysis for three months or longer
* Currently on a phosphate binder(s)
* Considered compliant with phosphate binders and hemodialysis therapy
* Willing to avoid any intentional changes in diet such as fasting or dieting
* Have the following documented local laboratory measurements:a.Two most recent consecutive serum phosphorus measurements that are ≥ 3.0 and ≤ 6.5 (6.5) mg/dL within 60 days of screening; b.A most recent intact parathyroid hormone (iPTH) measurement ≤ 800 pg/mL within 90 days of screening
* Have the following central laboratory measurements: a.A serum phosphorus measurement > 5.5 mg/dL at randomization (Week 0);b.A serum iPTH measurement ≤ 800 pg/mL at screening
* Have not participated in any other investigational drug studies within 30 days prior to enrollment
* Level of understanding and willingness to cooperate with all visits and procedures as described by the study personnel
* Willing and able to take sevelamer alone as a phosphate binder for the duration of the study
* Willing and able to maintain screening doses of lipid medication for the duration of the study, except for safety reasons
* Willing and able to avoid antacids and phosphate binders containing aluminum, magnesium, calcium or lanthanum for the duration of the study unless prescribed as an evening calcium supplement
* If female and of childbearing potential (pre-menopausal and not surgically sterile), willing to use an effective contraceptive method throughout the study, which includes barrier methods, hormones, or intrauterine devices (IUDs)
* Life expectancy of 12 months or greater
* Willing and able to provide informed consent

Exclusion Criteria:

* Active bowel obstruction, dysphagia, swallowing disorder, or severe gastrointestinal (GI) motility disorders
* Active ethanol or drug abuse, excluding tobacco use
* In the opinion of the Investigator, subject has poorly controlled diabetes mellitus, poorly controlled hypertension, active vasculitis, HIV infection, or any clinically significant unstable medical condition
* Use of anti-arrhythmic or anti-seizure medications for the use of arrhythmia or seizure disorders
* Known hypersensitivity to sevelamer or any constituents of the study drug
* Pregnant or breast-feeding
* Evidence of active malignancy except for basal cell carcinoma of the skin
* Unable to comply with the requirements of the study
* Any other condition which, in the opinion of the Investigator, will prohibit the subject's inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2006-01; Primary Completion 2007-03 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Demonstrate the efficacy of sevelamer carbonate powder dosed QD with the largest meal to sevelamer hydrochloride tablets dosed TID with meals on the control of serum phosphorus | Up to 24 weeks
Evaluate the safety and tolerability of sevelamer carbonate powder dosed QD with the largest meal compared to sevelamer hydrochloride tablets dosed TID with meals | Up to 24 weeks

SECONDARY OUTCOMES:
Compare sevelamer carbonate powder dosed QD with the largest meal to sevelamer hydrochloride tablets TID with meals on serum calcium-phosphorus product and serum lipid profile | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (29):
- United States (29):
  - Clinical Research Center, Birmingham, Alabama
  - Gadsden Dialysis, Gadsden, Alabama
  - Holy Cross Renal Care, Mission Hills, California
  - Nephrology Educational Services and Research, Tarzana, California
  - Crystal Rivers Dialysis Center, Crystal River, Florida
  - Outcomes Research International, Inc., Hudson, Florida
  - Central Dialysis Center, Atlanta, Georgia
  - Atlanta Nephrology Referral Center, Decatur, Georgia
  - FMC Marietta, Marietta, Georgia
  - Horizon Healthcare Associates, Flossmoor, Illinois
  - Indiana University Hospital, Indianapolis, Indiana
  - Ochsner Clinic Foundation, Nephrology Research, New Orleans, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - Southwest Mississippi Nephrology, PLLC, Brookhaven, Mississippi
  - Nephrology Associates, P.C., Columbus, Mississippi
  - Nephrology & Hypertension Associates, LTD, Tupelo, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Hypertension and Nephrology Associates, Eatontown, New Jersey
  - Winthrop University Dialysis Center, Mineola, New York
  - Davita, The Bronx, New York
  - Kidney and Hypertension Center, Cincinnati, Ohio
  - Renal Care Group, Cleveland, Ohio
  - Lewiston Dialysis Center, Lewistown, Pennsylvania
  - Medical Nephrology Associates, Dyersburg, Tennessee
  - Nephrology Associates, P.C., Nashville, Tennessee
  - Renal Research Inc. at the Kidney Institute, Houston, Texas
  - Gambro Healthcare - Charlottesville, Charlottesville, Virginia
  - Clinical Research of Tidewater, Norfolk, Virginia
  - Virginia Commonwealth University, Division of Nephrology, Richmond, Virginia